CLINICAL TRIAL: NCT04778943
Title: Oblique Lateral Interbody Fusion Versus Minimally Invasive Transforaminal Lumbar Interbody Fusion for Lumbar Spinal Stenosis
Brief Title: Oblique Lateral Interbody Fusion Versus Minimally Invasive Transforaminal Lumbar Interbody Fusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Fei-Long Wei, Clinical Professor, Tang-Du Hospital
Other Study IDs: TDGKJZ
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; OLIF; MIS-TLIF; postoperative improvements
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oblique lateral interbody fusion (OLIF): Patients with lumbar spinal stenosis undergoing oblique lateral interbody fusion (OLIF)
  Interventions: Other: Surgery(OLIF and MIS-TLIF)
- minimally invasive transforaminal lumbar interbody fusion (MIS-TLIF): Patients with lumbar spinal stenosis undergoing minimally invasive transforaminal lumbar interbody fusion (MIS-TLIF)
  Interventions: Other: Surgery(OLIF and MIS-TLIF)

INTERVENTIONS:
Other: Surgery(OLIF and MIS-TLIF) — oblique lateral interbody fusion (OLIF); minimally invasive transforaminal lumbar interbody fusion (MIS-TLIF)

SUMMARY:
The investigators will retrospectively study lumbar spinal stenosis patients who underwent OLIF or MIS-TLIF with percutaneous pedicle screw fixation between January 2016 and December 2019.The investigators will measure estimated blood loss, operative time, hospital stay, cost, reoperation, and complication incidence, visual analogue scale (VAS), Oswestry Disability Index (ODI), Japanese Orthopaedic Association (JOA), and Short Form-36 (SF-36) scores, discal and foraminal height, lumbar lordotic angle, and fusion status.The investigators will conduct to evaluate postoperative improvements, complications, and reoperation rates between patients with lumbar spinal stenosis (LSS) undergoing oblique lateral interbody fusion (OLIF) or minimally invasive transforaminal lumbar interbody fusion (MIS-TLIF).

ELIGIBILITY:
Inclusion Criteria:

* LSS due to neurogenic claudication; Central stenosis or lateral stenosis who need surgery; Single-level, low-grade (Meyerding grade 1 or 2) isthmic spondylolisthesis or degenerative spondylolisthesis; and imaging findings consistent with the symptoms of LSS.

Exclusion Criteria:

* trauma, active infection, malignant tumors, spinal deformity, previous lumbar fusion, multi-segment fusion, multi-level, high-grade (Meyerding grade 3 or 4) isthmic spondylolisthesis or degenerative spondylolisthesis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with LSS and underwent either MIS-TLIF or OLIF surgery between January 2016 and December 2019.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-02-28 (Estimated); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-03-29 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI), , and Short Form-36 (SF-36) scores; discal and foraminal height; lumbar lordotic angle; and fusion status. | 2 Years
  Before surgery and at the last follow-up, the following information was recorded

SECONDARY OUTCOMES:
Japanese Orthopaedic Association (JOA) | 2 Years
  Before surgery and at the last follow-up, the following information was recorded
visual analogue scale (VAS) | 2 Years
  Before surgery and at the last follow-up, the following information was recorded
Short Form-36 (SF-36) scores | 2 Years
  Before surgery and at the last follow-up, the following information was recorded
Major Complication rate | 2 Years

IPD SHARING:
Plan to Share IPD: Undecided